CLINICAL TRIAL: NCT05530070
Title: Cardiovascular Risk Factors in Coeliac Disease: a Series of Studies
Acronym: ARCTIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pecs (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 27521-5/2022/EÜIG
Record Dates: First submitted 2022-08-03; First posted 2022-09-07 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-05

CONDITIONS: Coeliac Disease
Keywords: coeliac disease; cardiovascular risk; body composition; dietary intervention
MeSH Terms: conditions — Celiac Disease | interventions — Diet Therapy; Standard of Care

STUDY DESIGN:
Intervention Model Description: This trial is a series of three multicentric studies. It includes 1) a case-control study, which compares newly diagnosed CD patients (n=37) and CD patients on a GFD (n=99) to matched non-coeliac control subjects (n=136); 2) a prospective cohort study, which investigates how the outcomes change during a 1-year GFD started after diagnosis of CD (n=236); 3) an RCT, which investigates how a dietetic intervention (n=95) influences the outcomes, compared to standard of care (n=95), in CD patients following a strict GFD for at least 1 year. There will be no intervention for the sake of the study in the case-control and the cohort study. Parameters of interest will be assessed only once in the case-control study and twice in the cohort study. In the RCT, randomization will be carried out after the baseline dietary education and interview, in 1:1 allocation ratio. Parameters will be recorded at baseline and the end of the study.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Due to the nature of the study, the blinding of the participants is not possible. The blinding of the physicians, data managers and statisticians will be secured.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary intervention (Active Comparator): Patients randomized to the dietary intervention group.
  Interventions: Other: Dietary intervention; Diagnostic Test: Cardiovascular risk-related parameters
- Standard of care (Active Comparator): Patients randomized to the standard of care group.
  Interventions: Other: Standard of care; Diagnostic Test: Cardiovascular risk-related parameters

INTERVENTIONS:
Other: Dietary intervention — Patients will participate in a structured, group-based dietary counseling. Consultations will be organized online (Zoom meeting) lasting approximately 60 min/occasion. The intervention will include 6 sessions for 1 year (monthly for 5 months and finally at month 9). The aim of the counseling is to maintain a GFD and to develop a healthy lifestyle, in line with the Mediterranean diet.
  Arms: Dietary intervention
Other: Standard of care — Patients will receive standard of care and baseline dietary education.
  Arms: Standard of care
Diagnostic Test: Cardiovascular risk-related parameters — Anthropometric measurements (body height, body composition assessment-InBody 770), questionnaires (symptoms, quality of life, dietary adherence, diet quality, cardiovascular risk), assessment of sarcopenia (handgrip dynamometer), urine collection (dietary adherence - urine gluten immunogenic peptide detection), blood collection (immunological tests, hormone levels complemented with routine laboratory panel), transabdominal US examination to assess the extent of fatty liver disease.

SUMMARY:
This investigation examines the most important cardiovascular risk factors (e.g., metabolic parameters, body composition) and their changes in coeliac disease. The series of studies allow to assess body composition and cardiovascular risk-related metabolic parameters of newly diagnosed and treated coeliac patients in their complexity and to test if they change during therapy. The interventional part of the investigation aims to answer the question if a dietary intervention mitigates the unfavorable effects of unbalanced diet.

DETAILED DESCRIPTION:
The global prevalence of coeliac disease (CD) is increasing, which contributes to the disease's significant public health care burden. Body composition and metabolic parameters of coeliac patients differ from the healthy population. Patients with non-classical CD are not necessarily lean; they usually have normal body weight but can be even overweight or obese. In coeliac patients, bodyweight tends to elevate, whereas the body composition changes unfavourably during a gluten-free diet (GFD). A reason for gaining weight is the improvement of malabsorption but an important contributor is the nutrient composition of the GFD, which generally has a high calorie density with high carbohydrate and fat content while being low in fibre. While terminating or mitigating the inflammatory process - if done without adequate dietary control - a GFD can readily lead to weight gain and unfavourably metabolic consequences (e.g., dyslipidemia, fatty liver disease, insulin resistance). The result can be an increase in cardiovascular risk in CD patients with a normal or high body weight at diagnosis. However, limited information is available on the cardiovascular (CV) risk in coeliac disease, and the data are controversial. This study examines the body composition and cardiovascular risk-related metabolic parameters at the diagnosis and on a gluten-free diet in a Hungarian cohort of CD patients. The randomised controlled trial (RCT) investigates the effect of structured, repeated, group-based dietary education on the examined metabolic parameters and body composition.

This study aims to draw attention to a new aspect of the management of CD patients: from a metabolic and cardiovascular point of view. Findings will help to identify which parameters are beneficial to optimize and re-assess during follow-up in CD.

ELIGIBILITY:
Inclusion Criteria (applies to all subjects):

* Age should be over 18 years.
* Blood collection must be indicated with medical conditions.
* Signed informed consent.

Inclusion Criteria (applies to specific cohorts of patients):

* The diagnosis of CD should be set up according to the current guidelines (based on serology and histology in adults or as per the European Society for Paediatric Gastroenterology Hepatology and Nutrition (ESPGHAN) guideline in children).
* The newly diagnosed CD patients should be on a gluten-containing diet.
* Patients following a GFD for at least 1 year should exhibit good dietary adherence.
* In the randomized controlled trial (RCT), strict dietary adherence will be established based on CD-specific serology (normal level of antibodies), urine gluten immunogenic peptides (negative urine test), and dietary interview (convincing knowledge on the GFD and positive attitude towards strict adherence). Adherence to the mediterranean diet should be suboptimal (≤ 8 Medietrranean Diet Score). RCT-patients must have internet access and must be capable to attend the online sessions for 1 year.
* Control subjects should be free from CD according to the recent guidelines and should be on a gluten-containing diet.

Exclusion Criteria:

* Chronic conditions:

  * Estimated glomerular filtration rate calculated with the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula is <60mL/min/1.73m2 (CKD3 or more severe kidney failure).
  * Liver cirrhosis in Child-Pugh class B-C.
  * Heart failure (New York Heart Association (NYHA) III-IV).
  * Active malignant diseases.
* Any acute diseases or acute deterioration of underlying chronic conditions.
* Diseases that may be associated with clinically relevant malabsorption.
* Refractory CD.
* Pregnancy, lactation.
* Patients unable to understand the essentials of the informed consent.
* Lack of consent or withdrawal of consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Percent body fat | 1 year
  Percent body fat in percentage measured by an InBody 770 body composition analyzer.

SECONDARY OUTCOMES:
Waist circumference | 1 year
  CV risk assessment will be performed by measuring waist circumference in centimeters.
Blood pressure | 1 year
  CV risk assessment will be performed by measuring blood pressure in Hgmm.
Fatty liver disease | 1 year
  Transabdominal ultrasonography will be used to assess the extent of fatty liver disease (based on non-alcoholic fatty liver disease-liver fat score (NAFLD-LFS), with a score range of 0-3).
Cardiovascular risk assessment | 1 year
  CV risk assessment will be performed by the Systematic Coronary Risk Evaluation (SCORE) chart.
Coeliac disease-related symptoms | 1 year
  CD-related symptoms will be assessed by the Celiac Symptom Index (CSI).
Coeliac disease-specific quality of life | 1 year
  CD-specific quality of life questionnaire will be also used (Celiac Disease Quality of Life (CD-QoL).
Disease activity | 1 year
  Disease activity will be estimated by tissue transglutaminase (tTG) levels.
Sarcopenia | 1 year
  Sarcopenia will be assessed based on body composition and handgrip strength via handgrip dynamometer.
Triglyceride level | 1 year
  Triglyceride level in mmol/L.
Cholesterol level | 1 year
  Cholesterol (total, HDL and LDL lipoproteins) level in mmol/L.
Fasting glucose level | 1 year
  Fasting glucose level in mmol/L.
Fasting insulin level | 1 year
  Fasting insulin level in mmol/L.
Haemoglobin (Hb) A1c level | 1 year
  HbA1c level in percentage.
Homeostasis Model Assessment (HOMA) index | 1 year
  HOMA index
Bilirubin level | 1 year
  Bilirubin level in µmol/L.
Uric acid level | 1 year
  Uric acid µmol/L.
Urea level | 1 year
  Urea level in mmol/L.
Creatinine level | 1 year
  Creatinine level in µmol/L.
Sodium level | 1 year
  Sodium level in mmol/L.
Potassium level | 1 year
  Potassium level in mmol/L.
Calcium level | 1 year
  Calcium level in mmol/L.
Vitamin D | 1 year
  Vitamin D level in ng/mL.
Vitamin B12 | 1 year
  Vitamin B12 level in pg/mL.
Folic acid level | 1 year
  Folic acid level in µg/L.
Iron level | 1 year
  Iron level in µmol/L.
Ferritin level | 1 year
  Ferritin level in µg/L.
Transferrin level | 1 year
  Transferrin level in g/L.
Transferrin saturation | 1 year
  Transferrin saturation in percentage.
International Normalized Ratio (INR) | 1 year
  INR
Aspartate aminotransferase level | 1 year
  Aspartate aminotransferase level in U/L.
Alanine aminotransferase level | 1 year
  Alanine aminotransferase in U/L.
Fibrosis-4 (FIB-4) Index | 1 year
  FIB-4 Index for liver fibrosis.
Total protein level | 1 year
  Total protein level in g/L.
Albumin level | 1 year
  Albumin level in g/L.
Immunoglobulins | 1 year
  Immunoglobulins in U/mL.
High-sensitivity C-reactive protein (hs-CRP) level | 1 year
  hs-CRP level in mg/L.
Fibrinogen level | 1 year
  Fibrinogen level in g/L.
Blood counts | 1 year
  Blood counts in Giga/L.
Homocysteine levels | 1 year
  Homocysteine levels in µmol/L.
Interleukin-6 levels | 1 year
  Interleukin-6 levels in ng/L.
Leptin levels | 1 year
  Leptin levels in ng/mL.
Ghrelin levels | 1 year
  Ghrelin levels in pg/mL.
Adiponectin levels | 1 year
  Adiponectin levels in µg/mL.
Galectin-3 levels | 1 year
  Galectin-3 levels in ng/mL.
Dietary interview | 1 year
  Dietary adherence will be determined by dietary interview provided by an expertise dietitian.
Celiac Disease Adherence Test | 1 year
  Dietary adherence will be determined by the Celiac Disease Adherence Test (CDAT).
Coeliac-specific antibodies | 1 year
  Dietary adherence will be determined by coeliac-specific antibodies (tissue transglutaminase (tTG) immunoglobulin (Ig) A/IgG and endomysium antibody levels (EMA) IgA) in U/mL.
Urine gluten immunogenic peptide | 1 year
  Dietary adherence will be determined by urine gluten immunogenic peptide (GIP) measurement.
Diet composition | 1 year
  The composition of a GFD will be evaluated with the indicator of adherence to the Mediterranean diet, the Mediterranean Diet Score (MDS).
Body height | 1 year
  Height in centimeters measured by a stadiometer.
Body weight | 1 year
  Weight in kilograms measured by an InBody 770 body composition analyzer.
Body mass index | 1 year
  Body mass index in kg/m2 calculated by an InBody 770 body composition analyzer.
Body fat mass | 1 year
  Body fat mass in kilograms measured by an InBody 770 body composition analyzer.
Skeletal muscle mass | 1 year
  Skeletal muscle mass in kilograms measured by an InBody 770 body composition analyzer.
Visceral fat area | 1 year
  Visceral fat area in cm2 measured by an InBody 770 body composition analyzer.
Total body water | 1 year
  Total body water in liters measured by an InBody 770 body composition analyzer.

CONTACTS AND LOCATIONS:
Overall Officials: Judit Bajor, MD, PhD, Principal Investigator — Division of Gastroenterology, First Department of Medicine, University of Pécs, 7624 Pécs, Hungary
Locations (1):
- First Department of Medicine, Medical School, University of Pécs, Pécs, Baranya, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Capristo E, Addolorato G, Mingrone G, De Gaetano A, Greco AV, Tataranni PA, Gasbarrini G. Changes in body composition, substrate oxidation, and resting metabolic rate in adult celiac disease patients after a 1-y gluten-free diet treatment. Am J Clin Nutr. 2000 Jul;72(1):76-81. doi: 10.1093/ajcn/72.1.76. PMID 10871564
- [Background] Newnham ED, Shepherd SJ, Strauss BJ, Hosking P, Gibson PR. Adherence to the gluten-free diet can achieve the therapeutic goals in almost all patients with coeliac disease: A 5-year longitudinal study from diagnosis. J Gastroenterol Hepatol. 2016 Feb;31(2):342-9. doi: 10.1111/jgh.13060. PMID 26212198
- [Background] Nunes-Silva JG, Nunes VS, Schwartz RP, Mlss Trecco S, Evazian D, Correa-Giannella ML, Nery M, Queiroz MS. Impact of type 1 diabetes mellitus and celiac disease on nutrition and quality of life. Nutr Diabetes. 2017 Jan 9;7(1):e239. doi: 10.1038/nutd.2016.43. PMID 28067892
- [Background] Villanueva M, Oyarzun A, Leyton B, Gonzalez M, Navarro E, Canales P, Ossa C, Munoz MP, Bascunan KA, Araya M. Changes in Age at Diagnosis and Nutritional Course of Celiac Disease in the Last Two Decades. Nutrients. 2020 Jan 6;12(1):156. doi: 10.3390/nu12010156. PMID 31935859
- [Background] Melini V, Melini F. Gluten-Free Diet: Gaps and Needs for a Healthier Diet. Nutrients. 2019 Jan 15;11(1):170. doi: 10.3390/nu11010170. PMID 30650530
- [Background] Costa A, Brito GAP. Anthropometric Parameters in Celiac Disease: A Review on the Different Evaluation Methods and Disease Effects. J Nutr Metab. 2019 Sep 9;2019:4586963. doi: 10.1155/2019/4586963. eCollection 2019. PMID 31583132
- [Background] Tucker E, Rostami K, Prabhakaran S, Al Dulaimi D. Patients with coeliac disease are increasingly overweight or obese on presentation. J Gastrointestin Liver Dis. 2012 Mar;21(1):11-5. PMID 22457854
- [Background] Suarez-Gonzalez M, Bousono Garcia C, Jimenez Trevino S, Iglesias Cabo T, Diaz Martin JJ. Influence of nutrition education in paediatric coeliac disease: impact of the role of the registered dietitian: a prospective, single-arm intervention study. J Hum Nutr Diet. 2020 Dec;33(6):775-785. doi: 10.1111/jhn.12800. Epub 2020 Aug 12. PMID 32790023
- [Background] Marciniak M, Szymczak-Tomczak A, Mahadea D, Eder P, Dobrowolska A, Krela-Kazmierczak I. Multidimensional Disadvantages of a Gluten-Free Diet in Celiac Disease: A Narrative Review. Nutrients. 2021 Feb 16;13(2):643. doi: 10.3390/nu13020643. PMID 33669442
- [Derived] Vereczkei Z, Szakacs Z, Peresztegi MZ, Lemes K, Hagymasi K, Dako S, Dako E, Lada S, Faluhelyi N, Szekeres G, Pasztor G, Farkas N, Par G, Mezosi E, Bajor J. Influence of a structured, 1-year-long dietary intervention regarding body composition and cardiovascular risk (ARCTIC) in coeliac disease: a protocol of a multicentre randomised controlled trial. BMJ Open. 2024 Oct 8;14(10):e084365. doi: 10.1136/bmjopen-2024-084365. PMID 39384235
- [Derived] Vereczkei Z, Imrei M, Szakacs Z, Kovari B, Papp V, Lenart Z, Berki T, Szirmay B, Farkas N, Balasko M, Habon T, Hegyi P, Bajor J. Cardiovascular risk factors in coeliac disease (ARCTIC): a protocol of multicentre series of studies. BMJ Open. 2023 Sep 13;13(9):e068989. doi: 10.1136/bmjopen-2022-068989. PMID 37709338